CLINICAL TRIAL: NCT06152107
Title: A Multi-center, Randomized Controlled Study to Evaluate the Efficacy and Safety of Precise Subsegmental Treatment With InterVapor for Severe Emphysema
Brief Title: A Multi-center RCT to Evaluate Subsegmental BTVA Treatment for Severe Emphysema
Acronym: BTVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IS23073
Record Dates: First submitted 2023-11-16; First posted 2023-11-30 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Severe Emphysema
Keywords: Bronchoscopic Thermal Vapor Ablation (BTVA); Chronic obstructive pulmonary disease (COPD); Severe emphysema; Bronchoscopic lung volume reduction (BLVR)
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subsegmental BTVA treatment plus optimal medical therapy (GOLD guidelines) (Experimental): Patients in experimental group will be treated with the InterVapor System in at least 2 subsegments of different segments(unless the two most severe subsegments are located in the same segment) per single procedure.
  Interventions: Procedure: BTVA treatment plus optimal medical therapy (GOLD guidelines)
- segmental BTVA treatment plus optimal medical therapy (GOLD guidelines) (Active Comparator): Patients in control group will be treated with the InterVapor System in at least 1 segment per single procedure.
  Interventions: Procedure: BTVA treatment plus optimal medical therapy (GOLD guidelines)

INTERVENTIONS:
Procedure: BTVA treatment plus optimal medical therapy (GOLD guidelines) — Patients in experimental group will be treated with the InterVapor System in at least 2 subsegments of different segments(unless the two most severe subsegments are located in the same segment). Patients in control group will be treated with the InterVapor System in at least 1 segment.
  A sequential procedure allows for at least 6 weeks and no longer than 6 months after the first procedure. Patients in both groups will receive ipsilateral hemithorax treatment per procedure, with a treatment volume (air + tissue) of ≤1700 mL per procedure and ≥1000 mL cumulatively across two procedures. All patients will continue to receive optimal medical therapy (GOLD guidelines) for the duration of the study.
  Follow-up visits will be scheduled at 1, 3, 6 and 12 months following the second procedure with examination of pulmonary function tests, HRCT, 6-minute walk test, SGRQ-C, mMRC, CAT questionnaires. All adverse events during the study will be recorded.

SUMMARY:
To compare the efficacy and safety of subsegmental treatment and segmental treatment with InterVapor in patients with severe emphysema

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old;
2. Patients with severe emphysema and with at least two treatable subsegments and 1 treatable segment in the ipsilateral lung assessed by QCT;
3. Non-smoking for 2 months prior to study enrollment, and remain abstinent from smoking for the duration of the study;
4. 15%predicted≤FEV1≤50%predicted, TLC≥100% predicted, RV≥150% predicted (and RV/ TLC≥55%);
5. 6MWD >140 meters (patients with lower limb disability or motor dysfunction will be exempted from the test)
6. mMRC score≥2;
7. Arterial blood gas levels of: PaCO2≤55 mmHg; PaO2>50 mmHg on room air;
8. Mentally and physically able to cooperate with the study procedures and to provide informed consent prior to study enrollment.

Exclusion Criteria:

1. Contraindications to bronchoscopy, such as:

   Prior myocardial infarction within 1 month, unstable myocardial ischaemia, ejection fraction (EF) ≤ 40%; Active haemoptysis; Coagulation disorders; Malignant cardiac arrhythmia, severe pulmonary hypertension, extreme systemic failure, etc;
2. Concomitant illnesses or medications that would pose a significant increased risk for complications following treatment with InterVapor. Examples of particular relevance include: immune system disorders, immunosuppressant medications of clinical relevance, bleeding disorders and unstable cardiovascular conditions, history of asthma or alpha-1 antitrypsin deficiency;
3. Use of morphine derivatives within 4 weeks prior to screening;
4. Taking more than 10 mg prednisolone or equivalent daily glucocorticoids at the screening visit;
5. Recent COPD exacerbation in preceding 6 weeks;
6. Severe emphysema in both the upper and lower lobes of the contralateral lungs, defined as %LAA-950 assessed by HRCT as a percentage of whole lung lobe volume > 40%;
7. Presence of single large bulla (defined as > 1/3 volume of lobe) or a paraseptal distribution of emphysema in the target lobe;
8. Presence of active pathogen related infection or symptoms indicative of active infection (e.g. fever, elevated WBC, etc.);
9. History of heart and/or lung transplant, lung volume reduction surgery (LVRS), median sternotomy, bullectomy, thoracic surgery with removal of lung tissue and endobronchial lung volume reduction (via valves, coils, stents, etc.);
10. Highly suspicious malignant pulmonary nodules in the lungs as assessed by specialist;
11. Pregnant or breastfeeding;
12. Current enrollment in any other investigational study which has not completed requisite follow-up;
13. Any conditions assessed by investigator that make patients inappropriate for enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in FEV1 | 6 months following the second procedure
  Improvement in FEV1 between experimental group vs control group at 6 months following the second procedure

SECONDARY OUTCOMES:
Changes in lung volumes by HRCT | 6 and 12 months following the second procedure
  Changes in lung volumes from baseline as assessed by HRCT at 6,12 months
Changes in FEV1 | 12 months following the second procedure
  Changes in FEV1 from baseline at 12 months
Changes in Quality-of-Life score | 6 and 12 months following the second procedure
  Changes in Quality-of-Life score as assessed by the SGRQ-C questionnaire from baseline at 6,12 months
Changes in FVC | 6 and 12 months following the second procedure
  Changes in FVC from baseline at 6,12 months
Changes in RV | 6 and 12 months following the second procedure
  Changes in RV from baseline at 6,12 months: RV
Changes in TLC | 6 and 12 months following the second procedure
  Changes in TLC from baseline at 6,12 months
Changes in RV/TLC | 6 and 12 months following the second procedure
  Changes in RV/TLC from baseline at 6,12 months
Changes in DLCO | 6 and 12 months following the second procedure
  Changes in DLCO from baseline at 6,12 months
Changes in 6MWD | 6 and 12 months following the second procedure
  Changes in 6MWD from baseline at 6,12 months (patients with lower limb disability or motor dysfunction will be exempted from the test)
Changes in CAT | 6 and 12 months following the second procedure
  Changes in CAT from baseline at 6,12 months
Changes in mMRC | 6 and 12 months following the second procedure
  Changes in mMRC from baseline at 6,12 months
A binary responder rate analysis will be performed to determine Minimal Clinically Important Difference (MCID) | 6 and 12 months following the second procedure
  A binary responder rate analysis will be performed to determine Minimal Clinically Important Difference (MCID) at 6,12 months:
  %predicted FEV1≥12% difference from baseline SGRQ-C≥8 points difference from baseline 6MWD≥26m from baseline
Incidence of Adverse Events | during or within 12 months after the operation
  Adverse events related to the procedure during or within 12 months after the operation

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Emergency General Hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Linyi People's Hospital, Linyi
  - Jiangxi Provincial People's Hospital, Nanchang
  - Shanghai Chest Hospital, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Hebei Provincial People's Hospital, Shijiazhuang
  - Sir Run Run Shaw Hospital affiliated to Zhejiang University School of Medicine, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gompelmann D, Shah PL, Valipour A, Herth FJF. Bronchoscopic Thermal Vapor Ablation: Best Practice Recommendations from an Expert Panel on Endoscopic Lung Volume Reduction. Respiration. 2018;95(6):392-400. doi: 10.1159/000489815. Epub 2018 Jun 12. PMID 29895029
- [Background] Shah PL, Herth FJ, van Geffen WH, Deslee G, Slebos DJ. Lung volume reduction for emphysema. Lancet Respir Med. 2017 Feb;5(2):147-156. doi: 10.1016/S2213-2600(16)30221-1. Epub 2016 Sep 29. PMID 27693408
- [Background] Bandyopadhyay S, Henne E, Gupta A, Barry R, Snell G, Strange C, Herth FJ. Segmental approach to lung volume reduction therapy for emphysema patients. Respiration. 2015;89(1):76-81. doi: 10.1159/000369036. Epub 2014 Dec 6. PMID 25500669
- [Derived] Yang H, Chen S, Ye L, Herth FJ, Sun J. Study protocol for a multicentre, randomised controlled trial in China to evaluate the efficacy and safety of precise subsegmental bronchoscopic thermal vapour ablation treatment in severe emphysema. BMJ Open. 2025 Oct 9;15(10):e099367. doi: 10.1136/bmjopen-2025-099367. PMID 41067776